CLINICAL TRIAL: NCT00418808
Title: Analysis of Movements of Singletons and Infants of Multiple Fetus Pregnancy as a Predictor of Developmental Delay
Brief Title: Early Movements as a Predictor of Future Developmental Delay
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4067-OB-CTIL
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2007-01-23 (Estimated); Status verified 2007-01

CONDITIONS: Cerebral Palsy; Premature Birth
Keywords: motor; development; multiple pregnancies; general movement; video recording
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
Cerebral Palsy (CP) is a major developmental problem. Major risk groups of CP, are preterm infants and multiple pregnancies. Previous studies using the General Movements methodology demonstrated early identification of CP, as early as 3 month of age. This method was implemented mainly on preterm infants this study goal is to enlarge the scope of the methodology to infants of multiple pregnancies. A second goal is to study early motor development and its future consequences by comparing the development of the infants of the same multiple pregnancy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a motor development problem with a prevalence of 2 per 1000 live birth. There are many etiologies to the syndrome such as: brain malformations, infections during pregnancy, pre and perinatal, anoxic brain damage etc. A high risk group for these causes is preterm infants and infants of multiple pregnancies.

Major motor deficits or brain insults are recognizable at early weeks but most of them are more subtle and are recognized at the age of one to two years. The General Movements methodology was developed by Prechtl HF is aimed to identify motor development deficits as early as 3 month. The methodology is using video recording to describe a trajectory of the development of spontaneous movements between birth and 3 month. Deviation from the trajectory was highly correlated with future motor mal-development.

In our work we will study the motor development of infants of multiple pregnancies. These infants are one of the risk groups to develop CP. We will use the General movements methodology to identify CP as early as possible. It will generalize its predicative power to this risk group. Moreover, we will enlarge our knowledge of motor development by comparing the development of infants of the same pregnancy.

ELIGIBILITY:
Inclusion Criteria for preterm infants:

* preterm infant under 37 weeks
* Normal or intraventricular hemorrhage grade I at U/S examination
* No neurological family history
* No maternal drug use with neurological effect during pregnancy
* Normal prenatal history such as: no evidence of hypoxic ischemic encephalopathy
* No convulsions
* Normal karyotype
* No major congenital heart defect
* Dizygotic twins

Inclusion Criteria for full term infants:

* Normal physiological examination
* No neurological family history
* No maternal drug use with neurological effect during pregnancy

Ages: 2 Days to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50
Dates: Start 2006-08; Study Completion 2009-08

CONTACTS AND LOCATIONS:
Overall Officials: Omer Bar-Yosef, Dr., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel Litwinsky, Israel